CLINICAL TRIAL: NCT03223246
Title: Medication Education for Dosing Safety
Acronym: MEDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Margaret Samuels-Kalow, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2017P001482
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Pain; Fever
MeSH Terms: conditions — Pain; Fever

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention)
- Additional teaching (Experimental)
  Interventions: Other: Additional teaching

INTERVENTIONS:
Other: Additional teaching — A brief safety intervention, combining a pictorial handout, dosing demonstration with dispensed syringe, and teach-back for confirmation of understanding.
  Arms: Additional teaching

SUMMARY:
Acetaminophen and ibuprofen are two of the most commonly used medication products among children <12 years old, and these medications are frequently prescribed for patients leaving the emergency department (ED), but previous studies have shown that parents often leave the ED unsure of how to safely dose these medications at home. This study will be a randomized controlled trial of a brief medication safety intervention, and examining parental knowledge and implementation of appropriate weight-based dosing.

ELIGIBILITY:
Inclusion Criteria:

* parents of children between ages of 90 days to 11.9 years
* being discharged with a plan for use of liquid acetaminophen (any age) or ibuprofen (limited to those >6 months old). The clinical team will determine planned medication use.
* parental fluency in English or Spanish
* ability to be reached by telephone over the next 7 days
* planned discharge home.

Exclusion Criteria:

* presence of a complex chronic condition in the child
* planned use of a non-standard weight-based medication dose.
* Families will also be excluded if the adult with the child is not a parent or legal guardian.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Samuels-Kalow, MD MSHP, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naureckas Li C, Camargo CA Jr, Faridi M, Espinola JA, Hayes BD, Porter S, Cohen A, Samuels-Kalow M. Medication Education for Dosing Safety: A Randomized Controlled Trial. Ann Emerg Med. 2020 Nov;76(5):637-645. doi: 10.1016/j.annemergmed.2020.07.007. Epub 2020 Aug 15. PMID 32807539

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Standard discharge care
Period: 48-72 Hours
Arm/Group | Usual Care | Additional Teaching
Started | 83 | 66
Completed | 62 | 35
Not Completed | 21 | 31
Period: 5-7 Days
Arm/Group | Usual Care | Additional Teaching
Started (Note: participants were called at 5-7 days even if they could not be reached at 48-72 hours) | 83 | 66
Completed | 41 | 35
Not Completed | 42 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Additional Teaching | Total
Number analyzed (Participants) | 83 | 66 | 149
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [29 to 39] | 34 [30 to 37] | 33 [30 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 54 | 115
  Male | 22 | 12 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic, White | 28 | 25 | 53
  Non-Hispanic, Black | 7 | 8 | 15
  Hispanic | 43 | 30 | 73
  Other | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 83 | 66 | 149
Health literacy (as measured by Newest Vital Sign) [Median (Inter-Quartile Range); unit: units on a scale] — Health literacy was measured by the Newest Vital Sign, which is scored from a minimum of 0 points to a maximum of 6 points. Higher scores represent higher health literacy.
  units on a scale | 4 [2 to 6] | 4 [2 to 6] | 4 [2 to 6]
Language of study administration [Count of Participants; unit: Participants]
  English | 59 | 51 | 110
  Spanish | 24 | 15 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Safe Dosing at 48-72 Hours
Description: Number of participants reporting dosing within 20% of the weight-based dose for the child at 48-72 hours
Time Frame: 48-72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Additional Teaching
Number analyzed (Participants) | 62 | 35
Participants | 28 | 25

2. Secondary Outcome: Number of Participants Reporting Persistence of Safe Dosing at 5-7 Days
Description: Number of participants reporting dosing within 20% of the weight-based dose for the child at 5-7 days
Time Frame: 5-7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Additional Teaching
Number analyzed (Participants) | 41 | 35
Participants | 22 | 26

3. Secondary Outcome: Number of Participants Reporting Contact With Other Providers at 48-72 Hours
Description: Number of participants reporting visit to primary care or emergency department providers at 48-72 hours
Time Frame: 48-72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Additional Teaching
Number analyzed (Participants) | 62 | 35
Participants | 29 | 18

4. Secondary Outcome: Number of Participants Reporting Contact With Other Providers at 5-7 Days
Description: Number of participants reporting visit to primary care or emergency department providers at 5-7 days.
Time Frame: 5-7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Additional Teaching
Number analyzed (Participants) | 41 | 35
Participants | 23 | 16

5. Other Pre Specified Outcome: Number of Participants Reporting Each Direction of Dosing Error at 48-72 Hours
Description: Number of participants reporting dosing error is above and/or below the weight-based dose for the child. Correct dosing was defined as 10mg/kg for ibuprofen and 10-15mg/kg for acetaminophen; dosing was considered incorrect if more than 20% above or below these values. Participants could be counted in more than one category for this outcome if they made more than one type of mistake (i.e. reported dose too high for acetaminophen and too low for ibuprofen).
Time Frame: 48-72 hours
Measure: Number; unit: participants
Arm/Group | Usual Care | Additional Teaching
Number analyzed (Participants) | 62 | 35
participants
  High | 9 | 4
  Low | 24 | 8
  Did not know dose | 9 | 1

6. Other Pre Specified Outcome: Number of Participants Reporting Each Direction of Dosing Error at 5-7 Days
Description: as for outcome 5
Time Frame: 5-7 days
Measure: Number; unit: participants
Arm/Group | Usual Care | Additional Teaching
Number analyzed (Participants) | 41 | 35
participants
  High | 6 | 3
  Low | 12 | 5
  Did not know dose | 2 | 1

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Usual Care | Additional Teaching
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/66
Serious Adverse Events (participants affected / at risk) | 2/83 | 2/66
Other Adverse Events (participants affected / at risk) | 16/83 | 19/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=83) | Additional Teaching (N=66)
Patient admitted (Social circumstances) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=83) | Additional Teaching (N=66)
Worsen at home (Social circumstances) | 16 (16) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT03223246/Prot_SAP_000.pdf